CLINICAL TRIAL: NCT02714062
Title: A Randomized, Double-Blind, Placebo-Controlled, Pharmacokinetic and Pharmacodynamic Study of VI-0521 in Obese Adolescents
Brief Title: A Pharmacokinetic Study Comparing VI-0521 With Placebo in Obese Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OB-402
Record Dates: First submitted 2016-03-08; First posted 2016-03-21 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Obesity; Childhood Obesity
Keywords: Adolescent Obesity; Childhood Obesity; Qsymia; Pharmacokinetics; VI-0521; Phentermine; Topiramate
MeSH Terms: conditions — Pediatric Obesity | interventions — Sugars; Qsymia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Days 1-56: Placebo
  Interventions: Drug: Placebo
- VI-0521 Mid Dose (Experimental): * Days 1-14: VI-0521 (Phentermine/Topiramate 3.75 mg/23 mg)
  * Days 15-56: VI-0521 (Phentermine/Topiramate 7.5 mg/46 mg)
  Interventions: Drug: VI-0521 Mid Dose
- VI-0521 Top Dose (Experimental): * Days 1-14: VI-0521 (Phentermine/Topiramate 3.75 mg/23 mg)
  * Days 15-28: VI-0521 (Phentermine/Topiramate 7.5 mg/46 mg)
  * Days 29-42: VI-0521 (Phentermine/Topiramate 11.25 mg/69 mg)
  * Days 43-56: VI-0521 (Phentermine/Topiramate 15 mg/92 mg)
  Interventions: Drug: VI-0521 Top Dose

INTERVENTIONS:
Drug: Placebo — po once daily
  Other Names: Sugar Pill
  Arms: Placebo
Drug: VI-0521 Mid Dose — po once daily
  Other Names: Phentermine/Topiramate
  Arms: VI-0521 Mid Dose
Drug: VI-0521 Top Dose — po once daily
  Other Names: Phentermine/Topiramate
  Arms: VI-0521 Top Dose

SUMMARY:
The primary objective of this study is to describe the pharmacokinetic profiles of VI-0521 in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Provide written assent (of study subject);
* Adolescent ≥12 and <18 years of age;
* Have a BMI ≥ the 95th percentile of BMI for age and gender;
* Female subjects must be using adequate contraception;
* Willing and able to comply with all study requirements

Exclusion Criteria:

* Condition or disease interfering with metabolism;
* Any medical treatment with insulin;
* Hyperthyroidism, or clinically significant hypothyroidism;
* Any history of bipolar disorder or psychosis, major depressive disorder, or history of suicidal behavior or ideation, or any use of antidepressant medications;
* Use of chronic systemic glucocorticoid or steroid therapy;
* History of any eating disorders;
* Any history of laxative abuse;
* Prior bariatric surgery;
* Any history of nephrolithiasis;
* Any history of epilepsy, or treatment with anti-seizure medications;
* Positive urine drug screen;
* Current smoker or smoking cessation within the previous 3 months of screening;
* Obesity of a known genetic or endocrine origin;
* Treatment with any over-the-counter or prescription weight loss drug, or attention-deficit/hyperactivity disorder (ADHD);
* Allergy or hypersensitivity to phentermine or topiramate or history of anaphylaxis to any drug;
* Use of any investigational medication or device for any indication or participation in a clinical study within 30 days prior to screening; or
* Any medical or surgical condition which would impair the ability of the subject to complete the study, compromise the quality of study data, or pose an unacceptable risk to the safety of the subject.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hsia, M.D., Principal Investigator — Pennington Biomedical Research
Locations (4):
- United States (4):
  - Research Facility, Baton Rouge, Louisiana
  - Research Facility, Marrero, Louisiana
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Started | 14 | 15 | 13
Completed | 13 | 14 | 10
Not Completed | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose | Total
Number analyzed (Participants) | 14 | 15 | 13 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.56) | 14.4 (1.30) | 14.3 (1.55) | 14.3 (1.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 9 | 26
  Male | 5 | 7 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 7 | 6 | 24
  White | 3 | 6 | 6 | 15
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 15 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Apparent Clearance (CL/F) of Phentermine and Topiramate
Description: A Bayesian analysis was performed to derive posterior Bayes individual pharmacokinetic (PK) parameters.
Time Frame: On Days 14, 28, 42, and 56
Population: PK samples were not collected for some patients due to withdrawal, or missed visits, etc. As a result, number analyzed for some visits is less than overall number analyzed.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 15 | 13
L/h
  Day 14 (Phentermine): number analyzed (Participants) | 14 | 11
  Day 14 (Phentermine) | 7.33 (1.63) | 7.04 (2.65)
  Day 28 (Phentermine): number analyzed (Participants) | 14 | 12
  Day 28 (Phentermine) | 7.33 (1.63) | 7.18 (2.57)
  Day 42 (Phentermine): number analyzed (Participants) | 14 | 11
  Day 42 (Phentermine) | 6.82 (1.69) | 6.49 (2.15)
  Day 56 (Phentermine): number analyzed (Participants) | 14 | 10
  Day 56 (Phentermine) | 6.82 (1.69) | 6.67 (2.18)
  Day 14 (Topiramate): number analyzed (Participants) | 14 | 11
  Day 14 (Topiramate) | 1.32 (0.333) | 1.25 (0.307)
  Day 28 (Topiramate): number analyzed (Participants) | 14 | 12
  Day 28 (Topiramate) | 1.32 (0.333) | 1.27 (0.300)
  Day 42 (Topiramate): number analyzed (Participants) | 14 | 11
  Day 42 (Topiramate) | 1.25 (0.291) | 1.20 (0.257)
  Day 56 (Topiramate): number analyzed (Participants) | 14 | 10
  Day 56 (Topiramate) | 1.25 (0.291) | 1.18 (0.265)

2. Primary Outcome: Apparent Volume of Distribution (Vc/F) of Phentermine and Topiramate
Description: A Bayesian analysis was performed to derive posterior Bayes individual PK parameters.
Time Frame: On Days 14, 28, 42, and 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 15 | 13
L
  Day 14 (Phentermine): number analyzed (Participants) | 14 | 11
  Day 14 (Phentermine) | 289 (80.4) | 289 (70.4)
  Day 28 (Phentermine): number analyzed (Participants) | 14 | 12
  Day 28 (Phentermine) | 287 (79.8) | 291 (69.6)
  Day 42 (Phentermine): number analyzed (Participants) | 14 | 11
  Day 42 (Phentermine) | 284 (79.3) | 298 (62.1)
  Day 56 (Phentermine): number analyzed (Participants) | 14 | 10
  Day 56 (Phentermine) | 281 (78.8) | 299 (64.6)
  Day 14 (Topiramate): number analyzed (Participants) | 14 | 11
  Day 14 (Topiramate) | 46.8 (17.7) | 46.1 (13.5)
  Day 28 (Topiramate): number analyzed (Participants) | 14 | 12
  Day 28 (Topiramate) | 46.2 (17.5) | 46.6 (13.5)
  Day 42 (Topiramate): number analyzed (Participants) | 14 | 11
  Day 42 (Topiramate) | 45.7 (17.3) | 48.2 (11.5)
  Day 56 (Topiramate): number analyzed (Participants) | 14 | 10
  Day 56 (Topiramate) | 45.2 (17.2) | 47.5 (12.3)

3. Primary Outcome: Area Under the Curve (AUC) of Phentermine
Description: A Bayesian analysis was performed to derive posterior Bayes individual PK parameters. AUC from time 0 to 24 hours under steady-state.
Time Frame: On Days 14, 28, 42, and 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 15 | 13
ng•h/mL
  Day 14 (Phentermine): number analyzed (Participants) | 14 | 11
  Day 14 (Phentermine) | 533 (109) | 600 (205)
  Day 28 (Phentermine): number analyzed (Participants) | 14 | 12
  Day 28 (Phentermine) | 1066 (218) | 1171 (403)
  Day 42 (Phentermine): number analyzed (Participants) | 14 | 11
  Day 42 (Phentermine) | 1154 (240) | 1902 (576)
  Day 56 (Phentermine): number analyzed (Participants) | 14 | 10
  Day 56 (Phentermine) | 1154 (240) | 2469 (775)

4. Primary Outcome: Maximum Concentration (Cmax) of Phentermine
Description: A Bayesian analysis was performed to derive posterior Bayes individual PK parameters.
Time Frame: On Days 14, 28, 42, and 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 15 | 13
ng/mL
  Day 14 (Phentermine): number analyzed (Participants) | 14 | 11
  Day 14 (Phentermine) | 27.6 (5.34) | 30.3 (9.61)
  Day 28 (Phentermine): number analyzed (Participants) | 14 | 12
  Day 28 (Phentermine) | 55.3 (10.7) | 59.3 (19.0)
  Day 42 (Phentermine): number analyzed (Participants) | 14 | 11
  Day 42 (Phentermine) | 59.0 (11.6) | 94.2 (25.9)
  Day 56 (Phentermine): number analyzed (Participants) | 14 | 10
  Day 56 (Phentermine) | 59.1 (11.6) | 123 (34.8)

5. Secondary Outcome: Weight Loss
Description: Mean percent weight change from baseline to Day 56
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: Percent weight change
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 13 | 15 | 12
Percent weight change | 1.14 (2.810) | -3.77 (2.446) | -4.99 (3.410)

6. Secondary Outcome: Change in Waist Circumference
Description: Mean change in waist circumference from baseline to Day 56
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 13 | 15 | 12
cm | 0.1 (4.17) | -2.6 (5.63) | -4.8 (4.91)

7. Secondary Outcome: Change in Blood Pressure
Description: Mean change in blood pressure from baseline to Day 56
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 14 | 15 | 13
mmHg
  Mean change in systolic BP: number analyzed (Participants) | 13 | 15 | 13
  Mean change in systolic BP | -6.0 (12.42) | -3.3 (10.24) | -3.8 (9.64)
  Mean change in diastolic BP: number analyzed (Participants) | 13 | 15 | 13
  Mean change in diastolic BP | -2.2 (7.53) | 3.5 (8.11) | 2.1 (6.10)

8. Secondary Outcome: Change in OGTT of Fasting and 2-hour Glucose
Description: Mean changes in glycemic parameters (OGTT of fasting and 2-hour glucose) from baseline to Day 56
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 14 | 15 | 13
mg/dL
  Mean Change in OGTT of Fasting Serum Glucose: number analyzed (Participants) | 13 | 14 | 10
  Mean Change in OGTT of Fasting Serum Glucose | -3.2 (11.66) | 0.6 (4.65) | -2.1 (9.64)
  Mean Change in OGTT of 2-Hour Serum Glucose: number analyzed (Participants) | 13 | 13 | 10
  Mean Change in OGTT of 2-Hour Serum Glucose | -1.2 (33.23) | -3.9 (31.96) | -9.3 (16.57)
  Mean Change in OGTT of Fasting Serum Insulin: number analyzed (Participants) | 13 | 14 | 10
  Mean Change in OGTT of Fasting Serum Insulin | 3.28 (25.463) | -10.92 (31.474) | -8.03 (6.500)
  Mean Change in OGTT of 2-Hour Serum Insulin: number analyzed (Participants) | 13 | 13 | 10
  Mean Change in OGTT of 2-Hour Serum Insulin | 11.45 (123.842) | -54.13 (176.897) | -92.99 (104.468)

9. Secondary Outcome: Change in Lipid Parameters
Description: Mean percent changes in lipid parameters, including total cholesterol, LDL-C, HDL-C and triglycerides (TG) from baseline to Day 56
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 14 | 15 | 13
Percent Change
  Mean Percent Change in TC: number analyzed (Participants) | 13 | 15 | 11
  Mean Percent Change in TC | 0.26 (9.154) | -6.10 (10.857) | -1.73 (14.103)
  Mean Percent Change in LDL-C: number analyzed (Participants) | 13 | 15 | 11
  Mean Percent Change in LDL-C | 2.89 (16.532) | -4.42 (13.567) | 8.99 (26.718)
  Mean Percent Change in HDL-C: number analyzed (Participants) | 13 | 15 | 11
  Mean Percent Change in HDL-C | -3.16 (20.539) | -6.62 (9.887) | -12.55 (14.248)
  Mean Percent Change in TG: number analyzed (Participants) | 13 | 15 | 11
  Mean Percent Change in TG | 7.54 (42.040) | 0.05 (58.326) | -8.05 (47.167)

10. Secondary Outcome: Change in Visual Analog Scale (VAS) Hunger Scores
Description: Mean change in visual analog scale (VAS) hunger scores from baseline to Day 56. VAS hunger score is measured using a 10.0 cm horizontal line. The left end of this line is defined by word descriptors "not at all hungry" and corresponds to a VAS hunger score of 0.0. The right end of this line is defined by word descriptors "extremely hungry all the time" and corresponds to a VAS hunger score of 10.0. Subjects were asked "Please mark with a perpendicular line on the scale how hungry you were overall during the past week:" to best describes their overall level of hunger during the past week. Research staff measure the distance between the "0.0 = not at all hungry" anchor and the mark made by the subject (length to the nearest tenth of a centimeter) to score the measure.
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 13 | 15 | 12
units on a scale | -0.48 (1.975) | -1.26 (2.030) | -3.28 (2.314)

11. Secondary Outcome: Change in Visual Analog Scale (VAS) Satiety Scores
Description: Mean change in visual analog scale (VAS) satiety scores from baseline to Day 56. VAS satiety score is measured using a 10.0 cm horizontal line. The left end of this line is defined by word descriptors "very satisfied" and corresponds to a VAS satiety score of 0.0. The right end of this line is defined by word descriptors "not all at satisfied" and corresponds to a VAS satiety score of 10.0. Subjects were asked "Please mark with a perpendicular line on the scale how satisfied you were after eating during the past week:" to evaluate how satisfied subjects are after eating during the past week. Research staff measure the distance between the "0.0 = very satisfied" anchor and the mark made by the subject (length to the nearest tenth of a centimeter) to score the measure.
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 13 | 15 | 12
units on a scale | -0.74 (2.164) | -0.65 (1.758) | 0.18 (2.221)

12. Primary Outcome: Area Under the Curve (AUC) of Topiramate
Description: as for outcome 3
Time Frame: On Days 14, 28, 42, and 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg•h/mL
Arm/Group | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 15 | 13
μg•h/mL
  Day 14 (Topiramate): number analyzed (Participants) | 14 | 11
  Day 14 (Topiramate) | 18.5 (4.49) | 19.4 (4.75)
  Day 28 (Topiramate): number analyzed (Participants) | 14 | 12
  Day 28 (Topiramate) | 37.0 (8.98) | 38.2 (9.33)
  Day 42 (Topiramate): number analyzed (Participants) | 14 | 11
  Day 42 (Topiramate) | 38.8 (8.90) | 60.1 (13.1)
  Day 56 (Topiramate): number analyzed (Participants) | 14 | 10
  Day 56 (Topiramate) | 38.8 (8.90) | 81.4 (17.9)

13. Primary Outcome: Maximum Concentration (Cmax) of Topiramate
Description: A Bayesian analysis was performed to derive posterior Bayes individual PK parameters.
Time Frame: On Days 14, 28, 42, and 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 15 | 13
μg/mL
  Day 14 (Topiramate): number analyzed (Participants) | 14 | 11
  Day 14 (Topiramate) | 0.917 (0.226) | 0.952 (0.236)
  Day 28 (Topiramate): number analyzed (Participants) | 14 | 12
  Day 28 (Topiramate) | 1.84 (0.454) | 1.88 (0.465)
  Day 42 (Topiramate): number analyzed (Participants) | 14 | 11
  Day 42 (Topiramate) | 1.92 (0.454) | 2.90 (0.594)
  Day 56 (Topiramate): number analyzed (Participants) | 14 | 10
  Day 56 (Topiramate) | 1.92 (0.456) | 3.93 (0.817)

14. Secondary Outcome: Change in HOMA-IR
Description: Mean changes in glycemic parameters (HOMA-IR) from baseline to Day 56
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 13 | 14 | 10
μIU/mL | 0.65 (7.298) | -2.46 (7.513) | -1.82 (1.444)

15. Secondary Outcome: Change in Whole Body Insulin Sensitivity Index (WBISI) (Matsuda)
Description: Mean changes in glycemic parameters [Whole Body Insulin Sensitivity Index (WBISI) (Matsuda)] from baseline to Day 56. The Oral Glucose Tolerance Test (OGTT) were performed at Baseline and Day 56 using 75 g oral glucose load; blood samples were obtained at baseline and at 2 hours post glucose load for evaluation of both glucose and insulin levels. Insulin Sensitivity was measured by obtaining glucose and insulin levels in a fasting state and at 2 hours after administration of oral glucose load. Matsuda index = 10,000/SQRT [glucose concentration (mg/dL) (fasting)*insulin concentration (uIU/mL) (fasting)*glucose concentration (mg/dL) (2 hours after glucose load)*insulin concentration (uIU/ mL) (2 hours after glucose load)], with higher numbers indicating better insulin sensitivity.
Time Frame: 56 days
Population: The number of subjects with values at both time points (Baseline and Day 56)
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
Number analyzed (Participants) | 13 | 13 | 10
Index | -0.19 (1.758) | 0.55 (1.226) | 2.13 (2.921)

ADVERSE EVENTS:
Groups:
- Placebo: Placebo: Placebo, po once daily
- VI-0521 Mid Dose: VI-0521 Mid Dose: phentermine 7.5 mg and topiramate 46 mg, po once daily
- VI-0521 Top Dose: VI-0521 Top Dose: phentermine 15 mg and topiramate 92 mg, po once daily
Arm/Group | Placebo | VI-0521 Mid Dose | VI-0521 Top Dose
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 1/13
Other Adverse Events (participants affected / at risk) | 7/14 | 6/15 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | VI-0521 Mid Dose (N=15) | VI-0521 Top Dose (N=13)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | VI-0521 Mid Dose (N=15) | VI-0521 Top Dose (N=13)
Headache (Nervous system disorders) | 3 | 2 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 1
Urine osmolarity increased (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may publish the result of the study 12 months or longer after termination of the study. The PI will provide the sponsor a copy of any proposed publication at least 30 days prior to submission for publication.